CLINICAL TRIAL: NCT02778425
Title: Partial Splenic Embolization Combined with Endoscopic Therapies and NSBB Decreases the Variceal Rebleeding Rate and Increases Recompensation Rate in Cirrhosis Patients with Hypersplenism: a Multicenter Randomized Controlled Trial
Brief Title: The Treatment of Hepatocirrhosis and Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanjing Gao (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Jinan Military General Hospital (Other)
Responsible Party: Sponsor-Investigator, Yanjing Gao, Vice presidengt of Department of Gastroenterology of Qilu Hospital, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201602-QILU
Record Dates: First submitted 2016-05-08; First posted 2016-05-19 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2021-09

CONDITIONS: Hepatic Cirrhosis; Portal Hypertension
Keywords: Partial splenic embolization; Hypersplenism; Thrombocytopenia; Portal hypertension; Gastroesophageal varices; Secondary prophylaxis; Endoscopic variceal ligation; Non-selective beta-blocker; hepatic recompensation
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Hypersplenism; Thrombocytopenia | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (7):
- Secondary prevention-1 (Experimental): Endoscopic therapy+ beta blockers
  Interventions: Procedure: Endoscopic therapy+ beta blockers
- Secondary prevention-2 (Experimental): Endoscopic therapy+ PSE+beta blockers
  Interventions: Procedure: Endoscopic therapy+ PSE+beta blockers
- Primary prevention-1 (Experimental): Beta blockers
  Interventions: Procedure: beta blockers
- Primary prevention-2 (Experimental): Endoscopic therapy
  Interventions: Procedure: Endoscopic therapy
- Primary prevention-3 (Experimental): Endoscopic therapy+ PSE
  Interventions: Procedure: Endoscopic therapy+ PSE
- Acute bleeding-1 (Experimental): Somatostatin+endoscopic therapy
  Interventions: Procedure: Somatostatin+Endoscopic therapy
- Acute bleeding-2 (Experimental): Somatostatin+endoscopic therapy+PSE
  Interventions: Procedure: Somatostatin+Endoscopic therapy+PSE

INTERVENTIONS:
Procedure: Endoscopic therapy+ beta blockers — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).A standard dose of NSBB (propranolol) was applied to patients according to the Baveno VI recommendations if there were no contraindications.
  Arms: Secondary prevention-1
Procedure: Endoscopic therapy+ PSE+beta blockers — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).A standard dose of NSBB (propranolol) was applied to patients according to the Baveno VI recommendations if there were no contraindications.Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Secondary prevention-2
Procedure: beta blockers — A standard dose of NSBB (propranolol) was applied to the primary prevention patients according to the Baveno VI recommendations if there were no contraindications.
  Arms: Primary prevention-1
Procedure: Endoscopic therapy — Endoscopic variceal ligation (EVL) is for the primary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).
  Arms: Primary prevention-2
Procedure: Endoscopic therapy+ PSE — Endoscopic variceal ligation (EVL) is for the primary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Primary prevention-3
Procedure: Somatostatin+Endoscopic therapy — The first dose of 250 was injected intravenously, followed by a continuous iv infusion of 250 for 3-5 days. Endoscopic variceal ligation (EVL) is for the acute bleeding of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).
  Arms: Acute bleeding-1
Procedure: Somatostatin+Endoscopic therapy+PSE — The first dose of 250 was injected intravenously, followed by a continuous iv infusion of 250 for 3-5 days. Endoscopic variceal ligation (EVL) is for the acute bleeding of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Acute bleeding-2

SUMMARY:
This study compare the efficiency of partial splenic embolization +endoscopical therapy with endoscopical therapy alone in gastroesophageal variceal haemorrhage accompanied with splenomegaly or hypersplenism of hepatocirrhosis and portal hypertension treatment.

DETAILED DESCRIPTION:
Endoscopic therapy is the mature treatment of gastroesophageal variceal haemorrhage and PSE is an effective method for treatment of the hypersplenism and portal hypertension. Existing researches show that endoscopic therapy + PSE is more effective than endoscopic therapy alone in prevention of esophageal varices bleeding recurrence in the patients with liver cirrhosis. However, there is few articles which proved long-term effectiveness of endoscopic therapy + PSE, it needs further research on this issue. This study compares the efficiency of partial splenic embolization +endoscopic therapy with endoscopic therapy alone in the treatment of gastroesophageal variceal haemorrhage accompanied with splenomegaly or hypersplenism in the patients with hepatocirrhosis and portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients who had recovered from an episode of VH or patients who had survived from acute VH and there was no bleeding for consecutive 5 days
* Patients with a diagnosis of liver cirrhosis and portal hypertension on clinical examination, laboratory test, and imaging or histological examination
* Patients with hypersplenism and thrombocytopenia (platelets < 100,000/µL).

Exclusion criteria :

* Previous therapy (splenectomy, PSE, EVL, tissue adhesive injection, or usage of (NSBB) to prevent rebleeding
* Bleeding from isolated gastric or ectopic varices
* Hepatocellular carcinoma or other malignant tumors
* Contraindications for the use of NSBBs, hepatic failure, and Child-Pugh class C with large amount ascites, or grade 3-5 hepatic encephalopathy, or prothrombin activity ≤ 40%
* Hepatic failure
* Contraindications for PSE
* Pregnancy and lactation
* Inability to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was variceal rebleeding | 2 years
  The rebleeding rate of the varices in the EP group will compared to that in the E group during the follow up.
The primary outcome was the hepatic recompensation rate based on Baveno VII criteria after 1-year follow-up. | 2 years
  The hepatic recompensation rate based on Baveno VII criteria in the EP group will compared to that in the E group during the follow-up. Hepatic recompensation is a comprehensive assessment index defined as meeting all of the following criteria simultaneously: (1)Etiological Control: Removal/suppression/cure of the primary cause of cirrhosis (e.g., hepatitis C virus elimination, sustained suppression of hepatitis B virus, and sustained abstinence from alcohol in alcoholic cirrhosis); (2)Symptomatic Resolution: Regression of ascites (discontinuation of diuretics), remission of hepatic encephalopathy (discontinuation of lactulose/rifaximin), and absence of recurrent variceal bleeding (for at least 12 months); (3)Improvement in Liver Function: Stable improvement in liver function tests (albumin, INR, bilirubin).
  Assessed via lab tests (HCV RNA, HBV DNA, albumin, INR, bilirubin) and clinical evaluation (ascites, encephalopathy, endoscopy). Reported as binary (Yes/No).

SECONDARY OUTCOMES:
The secondary endpoints were severe variceal recurrence and mortality during the 2-year follow-up | 2 years
  The recurrence rate of the varices in the EP group will compared to that in the E group during the follow up.
Changes of the peripheral blood cell counts including white blood cell, red blood cell, and platelate counts in both group during 2-years follow up. | 2 years
  The physiological parameters including white blood cell (*10^9/L), red blood cell (*10^12/L) and platelte(*10^12/L) will compared between the two groups.
The secondary endpoints were changes in Child-Pugh Score, MELD Score, and Physiological Parameters during the follow-up. | 2 years
  Changes in liver function (Child-Pugh score, MELD score) and physiological parameters (white blood cell count [*10^9/L], red blood cell count [*10^12/L], platelet count [*10^12/L], hemoglobin [g/dL], and coagulation parameters) will be assessed and compared during the 1-year follow-up between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital,Shandong Universty
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol
Time Frame: 2021.1
Access Criteria: Open Access
URL: https://doi.org/10.1007/s12072-021-10155-0

REFERENCES:
- [Derived] Wei M, Chen Y, Wang M, Li J, Zeng Y, Sun X, Zhang A, Liu X, Zhou T, Gao Y. Partial splenic embolization combined with endoscopic therapies and vasoconstrictive drugs reduces rebleeding in cirrhosis patients with acute variceal bleeding and hypersplenism: a multicenter randomized controlled trial. J Gastroenterol. 2023 Nov;58(11):1144-1153. doi: 10.1007/s00535-023-02027-1. Epub 2023 Jul 24. PMID 37486372
- [Derived] Sun X, Zhang A, Zhou T, Wang M, Chen Y, Zhou T, Chen X, Xiu A, Peng Z, Cheng B, Liu X, Gao Y. Partial splenic embolization combined with endoscopic therapies and NSBB decreases the variceal rebleeding rate in cirrhosis patients with hypersplenism: a multicenter randomized controlled trial. Hepatol Int. 2021 Jun;15(3):741-752. doi: 10.1007/s12072-021-10155-0. Epub 2021 Feb 27. PMID 33638769